CLINICAL TRIAL: NCT06450002
Title: Calf Muscle Contraction During Walking: a New Critical Preposition in Clinical Biomechanics: A Conceptual Study
Brief Title: Calf Muscle Contraction During Walking
Status: Completed | Type: Observational
Sponsor: Noha Khaled Shoukry (Other)
Responsible Party: Sponsor-Investigator, Noha Khaled Shoukry, lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: PTCairoUniversity
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Calf Muscle Pulled
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: physical therapy — Tens and Hot packs for 20 minutes, ultrasound for 5 minutes on the back and back exercise in form of bridging exercise and core stability exercise

SUMMARY:
Walking is the most familiar form of exercise, the calf muscle plays an important role in the stance phase of the normal gait cycle of gait. The relative contribution of the calf muscle to the total positive work of the lower extremities during walking is approximately 51% and 73% in the elderly and younger people respectively. This study will explore the different types of calf muscle activation during normal gait cycle based on the previous literature and will introduce a new proposition in the biomechanics of calf muscle contraction..Also, this study will address the role of this muscle during gait and the effects of calf muscle weakness on the lumbar spine.

DETAILED DESCRIPTION:
400 patients with a history of calf muscles' weakness throughout the last 3 years will be included in the study. The patients suffered from unresolved CLBP with radiculopathy contralateral to their calf muscle atrophy (i.e., an ipsilateral calf muscle weakness induces contralateral lumbar radiculopathy) that did not respond to physical therapy or any medication for long patients in an out-patient clinic in Egypt (2016 to 2022) are screened for calf muscle weakness secondry to ankle injury. Patients with lumbar disc herniation (confirmed by MRI) and radiculopathy contralateral to the calf muscle weakness are recruited to participate in this study A better understanding of the calf muscle contraction can provide a valuable insight into how the calf muscle works during walking, predict calf muscle injuries and develop specific exercise to enable the patients with calf muscle dysfunction. …………………………………………………………………………………………………………………

ELIGIBILITY:
Inclusion Criteria:

* The patients suffered from unresolved CLBP with radiculopathy contralateral to their calf muscle atrophy (i.e., an ipsilateral calf muscle weakness induces contralateral lumbar radiculopathy) that did not respond to physical therapy or any medication for long

Exclusion Criteria:

* any spinal deformity or previous spinal surgeries. Spinal tumors or fracture or presence of active infection in the lumbar spine. Cauda equine lesion, the presence of any comorbidities such as hypertension, DM, hyperlipidemia, obesity, and any autoimmune disease, history of patients who suffered from cancer, unexplained weight loss, immunosuppression, prolonged use of steroids, intravenous drug use, urinary tract infection, pain that is increased or unrelieved by rest, fever, significant trauma related to age, bladder or bowel incontinence, urinary retention (with overflow incontinence), saddle anesthesia, loss of anal sphincter tone, major motor weakness in lower extremities, fever, and vertebral tenderness

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with a history of calf muscles' weakness throughout the last 3 years patients in an out-patient clinic in Egypt (2016 to 2022) are screened for calf muscle weakness secondry to ankle injury. Patients with lumbar disc herniation (confirmed by MRI) and radiculopathy contralateral to the calf muscle weakness are recruited to participate in this study
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
length of the calf muscle | three months
  ultrasosnography and EMG are used to detect the length of the calf muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided